CLINICAL TRIAL: NCT00006233
Title: Phase II Trial of Non-Myeloablative Allogeneic Peripheral Blood Stem Cell (PBSC) Transplantation Using Fludarabine, Low-Dose TBI, and Post-Transplant Immunosuppression With Cyclosporine and Mycophenolate Mofetil (MMF) Followed by Donor Lymphocyte Infusion in Selected Patients With Metastatic Melanoma
Brief Title: Combination Chemotherapy, Total-Body Irradiation, Peripheral Stem Cell Transplantation, and Lymphocyte Infusion in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 1462.00; FHCRC-1462.00; NCI-G00-1841; CDR0000068157 (Registry Identifier: PDQ)
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Cyclosporine; fludarabine phosphate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: mycophenolate mofetil
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as fludarabine use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy. Sometimes the transplanted cells can reject the body's normal tissues. Donor lymphocytes that have been treated in the laboratory may prevent this.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy, total-body irradiation, peripheral stem cell transplantation, and lymphocyte infusion in treating patients who have stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate in patients with metastatic melanoma treated with nonmyeloablative allogeneic peripheral blood stem cell transplantation with fludarabine and total body irradiation, followed by cyclosporine and mycophenolate mofetil, followed by donor lymphocyte infusion.
* Determine the disease-free and overall survival of patients treated with this regimen.
* Determine the toxicity of this nonmyeloablative conditioning regimen in these patients.

OUTLINE: Patients receive a conditioning regimen comprising fludarabine IV on days -4 to -2 and total body irradiation on day 0. Allogeneic peripheral blood stem cells are infused on day 0.

Patients receive oral cyclosporine twice a day on days -3 to 35 and tapered until day 56 and oral mycophenolate mofetil 3 times a day on days 0-40.

Patients with mixed chimerism and no graft-versus-host disease on day 56 receive donor lymphocyte infusion (DLI) over 30 minutes on day 65 unless there is evidence of increasing donor chimerism. DLI may be repeated every 65 days for up to 4 doses.

Patients are followed weekly for 3 months, monthly for 6 months, every 6 months through year 2, and then annually through year 5.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV melanoma
* Partial response, minor response, or stable disease after no more than 2 regimens of chemotherapy, immunotherapy, or chemoimmunotherapy
* Bidimensionally measurable disease by palpation on clinical exam or radiographic imaging
* HLA genotypically identical sibling donor available

  * Not an identical twin
  * Age 12 to 74
* No ocular melanoma
* No active or untreated brain metastases or transmural gastrointestinal metastases

PATIENT CHARACTERISTICS:

Age:

* 18 to 64

Performance status:

* Karnofsky 80-100%

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* SGOT and SGPT less than 2 times ULN

Renal:

* Creatinine clearance at least 40 mL/min

Cardiovascular:

* LVEF at least 40% if history of congestive heart failure
* No uncontrolled hypertension

Pulmonary:

* DLCO at least 50% of predicted
* No continuous supplementary oxygen

Other:

* Not pregnant
* Fertile patients must use effective contraception during and for 1 year after study participation
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No concurrent growth factors during mycophenolate mofetil administration

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2000-01; Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A. Thompson, MD, Study Chair — Seattle Cancer Care Alliance
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States